CLINICAL TRIAL: NCT03244306
Title: Pediatric and Young Adult Leukemia Adoptive Therapy (PLAT)-04: A Phase 1 Feasibility and Safety Study of CD22-CAR T Cell Immunotherapy for CD22+ Leukemia and Lymphoma
Brief Title: A Phase 1 Study of CD22-CAR TCell Immunotherapy for CD22+ Leukemia and Lymphoma
Acronym: PLAT-04
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLAT-04
Record Dates: First submitted 2017-08-03; First posted 2017-08-09 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Leukemia
Keywords: leukemia; CD 22; CAR T cell; pediatric; young adult; chimeric antigen receptor
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous CD22-specific CAR T-cells expressing EGFRt (Experimental)
  Interventions: Biological: Patient-derived CD22-specific CAR T-cells also expressing an EGFRt

INTERVENTIONS:
Biological: Patient-derived CD22-specific CAR T-cells also expressing an EGFRt — Patient-derived CD22-specific chimeric antigen receptor T-cells expressing an EGFRt

SUMMARY:
Patients with relapsed or refractory leukemia often develop resistance to chemotherapy and some patients who relapse following CD19 directed therapy relapse with CD19 negative leukemia. For this reason, the investigators are attempting to use T-cells obtained directly from the patient, which can be genetically modified to express a chimeric antigen receptor (CAR) to CD22, a different protein from CD19, expressed on the surface of the leukemic cell in patients with CD22+ leukemia. The CAR enables the T-cell to recognize and kill the leukemic cell through the recognition of CD22, a protein expressed on the surface of the leukemic cell in patients with CD22+ leukemia. This is a Phase 1 study designed to determine the safety and feasibility of the CAR+ T - cells and the feasibility of making enough to treat patients with CD22+ leukemia.

ELIGIBILITY:
Inclusion Criteria:

* First 3 subjects: male and female subjects age ≥ 18 years and < 27 years
* Subsequent subjects: 12 months of age and <27 years of age at the time of study enrollment
* Disease status (one of the following):

  1. If post-allogeneic hematopoetic cell transplant (HCT): confirmed CD22+ leukemia recurrence, defined as ≥0.01% disease
  2. If Relapse/Refractory status with no prior history of allogeneic HCT, one of:

     * 2nd or grater marrow relapse, with or without extramedullary disease
     * 1st marrow relapse at end of 1st month of re-induction with marrow having ≥0.01% blasts by morphology and/or MPF
     * Primary Refractory, defined as >5% blasts by multi-parameter flow after ≥2 separate induction regimens
     * Subject has indication for HCT but is ineligible, inclusive of persistent minimal residual disease
  3. CD22+ Lymphoma refractory or relapsed with no known curative therapies available
* Asymptomatic from CNS involvement, if present, and have a reasonable expectation that disease burden can be controlled in the interval between enrollment and T-cell infusion. Subjects with significant neurologic deterioration will not be eligible for T-cell infusion until stabilized.
* Free from active GVHD and off immunosuppressive GVHD therapy for 4 weeks.
* Lansky or Karnofsky performance score of ≥50
* Life expectancy of >8 weeks
* Recovered from acute toxic effects of all prior chemotherapy, immunotherapy, and radiotherapy
* ≥7 days post last chemotherapy administration (excluding intrathecal or maintenance chemotherapy)
* ≥7 days post last systemic corticosteroid administration
* No prior virotherapy
* Adequate organ function
* Adequate laboratory values
* Patients of childbearing/fathering potential must agree to use highly effective contraception
* Signed a written consent

Exclusion Criteria:

* Presence of active clinically significant CNS dysfunction
* Pregnant or breastfeeding
* Unable to tolerate apheresis procedure, including placement of temporary apheresis line if required
* Presence of active malignancy other than CD22+ leukemia or lymphoma
* Presence of active severe infection
* Presence of any concurrent medical condition that would prevent the patient from undergoing protocol-based therapy
* Presence of primary immunodeficiency/bone marrow failure syndrome
* Unwilling to participate in 15-year follow-up period that is required if CAR T cell therapy is administered

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2035-07 (Estimated)

PRIMARY OUTCOMES:
The adverse events associated with one or multiple CAR T-cell product infusions will be assessed | 30 days
  The type, frequency, severity, and duration of adverse events will be summarized
The number of successfully and unsuccessfully manufactured and infused CAR T-cell products will be assessed | 28 days
  Proportion of products successfully manufactured and infused

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Summers, MD, Study Chair — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No